CLINICAL TRIAL: NCT02837484
Title: The NuTech Affinity™ Membrane Product Evaluation for the Treatment of Chondral Defects
Brief Title: NuTech Affinity™ for the Treatment of Chondral Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NuTech Medical, Inc (Industry)
Collaborators: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD2015-11-04
Record Dates: First submitted 2016-07-14; First posted 2016-07-19 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Chondral Lesions; Cartilage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NuTech Affinity™ Membrane (Other): Sharp dissection of the defect will be performed being careful not to violate the subchondral bone sparing the calcified cartilage layer. After hemostasis is reached, the defect will be treated with an Affinity™ patch stabilized with fibrin glue.
  Interventions: Other: NuTech Affinity™ Membrane

INTERVENTIONS:
Other: NuTech Affinity™ Membrane — NuTech Affinity™ Membrane is an aseptically produced hypothermically stored amniotic membrane patch.

SUMMARY:
This study was designed to evaluate the long term effectiveness of a product used in knee surgery called Affinity™ Membrane.

DETAILED DESCRIPTION:
This is a one-arm prospective, non-randomized, longitudinal study with up to 10 patients from one orthopaedic clinic in the United States. Patients will be treated with Affinity™ a hypothermically preserved amniotic membrane.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signature of the IRB (Institutional Review Board) approved Informed Consent
2. Male or female participants between the ages of 18-55
3. If female:

   1. Actively practicing a contraception method, or
   2. Practicing abstinence, or
   3. Surgically sterilized, or
   4. Postmenopausal
4. Pretreatment arthroscopic confirmation indicating one or two contained or uncontained lesion(s) and equal to an ICRS Grade 3a, 3b, 3c, 3d of the femoral condyle or trochlear groove and OCD (Osteohondritis dissecans) lesions (Grade 4a) with healed bone base, which is non-sclerotic and no loss of bone greater than 6mm measured from the surrounding subchondral plate. Original pretreatment arthroscopic confirmation indicates that one or two lesion(s) are equal to an ICRS (Internation Cartilage Repair Society) Grade 3a, 3b, 3c, 3d contained lesion(s) that is equivalent to an Outerbridge Grade III or IV (greater than 50% loss of articular cartilage).
5. Has peripheral cartilage debridement to healthy cartilage that results in a lesion (s) with an area of > or = 1cm ^2 and < or = 5 cm^2.
6. PCL (Posterior Cruciate Ligament), LCL (Lateral Collateral Ligament) and MCL (Medical Collateral Ligament) in the affected knee are stable and the ACL (Anterior Cruciate Ligament) is stable or can be stabilized as a concomitant procedure.
7. Ipsilateral knee compartment has intact menisci (or requires partial meniscectomy resulting in stable menisci). No less than 60 degrees meniscal volume retained.
8. The contralateral knee is asymptomatic, stable, and fully functional.
9. Must be physically and mentally willing and able to comply with post-operative rehabilitation and routinely scheduled clinical and radiographic visit through 24 months.
10. Alignment: Mechanical axis must be no more than 6 degrees from neutral.
11. Must be at least 3 months post previous surgery.

Exclusion Criteria:

1. Clinical and/or radiographic disease diagnosis of the indexed affected joint that Includes:

   1. Osteoarthritis or avascular necrosis,
   2. Rheumatoid arthritis, or history of septic or reactive arthritis,
   3. Gout or history of gout or pseudogout in the affected knee,
   4. Osteochondritis dissecans of the knee with significant bone loss (greater than 6 mm deep measured from the subchondral plate)
   5. Associated damage to the underlying subchondral bone requiring a bone graft
2. History of secondary arthropathies (i.e. sickle cell disease, hemochromatosis, or autoimmune disease).
3. Uncontrolled diabetes.
4. Displays a high surgical risk due to unstable cardiac and/or pulmonary disease.
5. Has HIV or other immunodeficient state including subjects on immunosuppressant therapies, or has significant illness (metastasis of any type) that decreases the probability of survival to the 2 year endpoint.
6. Is at substantial risk for the need of organ transplantation, such as renal insufficiency.
7. Is pregnant or breast-feeding.
8. Body mass index > 35.
9. Has bipolar articular cartilage involvement or kissing lesions of the ipsilateral compartment, described as tibial or patellar lesions in the same compartment with greater than ICRS Grade 2 chondrosis.
10. Is participating concurrently in another clinical trial, or has participated in a clinical trial within 30 days of surgery.
11. Is receiving prescription pain medication other than NSAIDs or acetaminophen for conditions unrelated to the index knee condition, chronic use of anticoagulants, or taking corticosteroids.
12. Has a neuromuscular, neurosensory, or musculoskeletal deficiency that limits the ability to perform objective functional assessment of either knee.
13. Active joint infection.
14. Prior total meniscectomy of either knee.
15. Radiographically has >5 degrees of malalignment as measured from the hip, knee and ankle mechanical axis.
16. Has received within the past three months intra-articular hyaluronic acid therapy or cortisone injections in the index knee.
17. Prior realignment surgery in the affected knee within the past 6 months.
18. Failed microfracture treatment performed less than 12-months before inclusion visit.
19. Is receiving workman's compensation or currently involved in litigation relating to the index knee.
20. Has history of alcoholism, medication, or intravenous drug abuse, psychosis, is a prisoner, has a personality disorder (s), poor motivation, emotional or intellectual issues that would likely make the subject unreliable for the study, or any combination of variables in the investigator's judgment that should exclude a potential subject.
21. Had or have an aneurysm clip implanted, intraocular foreign bodies (commonly seen in welders), subcutaneous metal shards (found in sheet metal workers), or some shrapnel; additionally no cardiac pacemaker, defibrillator, implanted neurostimulater (TENS implants) some prosthetic heart valve (especially mitral valve), cochlear implant or other hearing aide, or has a tendency of claustrophobia. Tattoos that may contain iron-based dyes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Objective cartilage repair measured by MRI scanning | 6 months, 12 months and 24 months
Change from baseline for VAS scores | 3 months, 6 months, 12 months 18 months, and 24 months
Change from baseline of pain and functions scores on KOOS questionaire | 3 months, 6 months, 12 months, 18 months and 24 months

SECONDARY OUTCOMES:
Changes in patient-reported outcomes (PRO) questionnaires from baseline including IKDC (International Knee Documentation Committee) | 3 months, 6 months, 12 months, 18 months and 24 months
Histological assessment of optional cartilage biopsies | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sam Tabet, MD, Principal Investigator — New Mexico Orthopaedic Associates
Locations (1):
- New Mexico Orthopaedics, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tabet SK, Kimmerling KA, Hale GJ, Munson NR, Mowry KC. Hypothermically Stored Amniotic Membrane for the Treatment of Cartilage Lesions: A Single-Arm Prospective Study with 2-Year Follow-Up. Cartilage. 2022 Jan-Mar;13(1):19476035211072213. doi: 10.1177/19476035211072213. PMID 35073769